CLINICAL TRIAL: NCT03915886
Title: A Double-blind, Placebo-controlled, Randomized, Single Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-64530440 in Healthy Japanese Male Subjects
Brief Title: A Study of JNJ-64530440 in Healthy Japanese Male Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped due to a strategic decision.
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108603; 64530440HEP1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- JNJ-0440 (Low Dose) or Placebo (Experimental): Participants will receive single oral dose (low) of JNJ-0440 or matching placebo under fed conditions. The dose will be escalated based on the preliminary safety data from the preceding cohort as per sponsor and investigator discretion.
  Interventions: Drug: JNJ-0440; Drug: Placebo
- JNJ-0440 (Medium Dose) or Placebo (Experimental): Participants will receive single oral dose (medium) of JNJ-0440 or matching placebo under fed conditions. The dose will be escalated based on the preliminary safety data from the preceding cohort as per sponsor and investigator discretion.
  Interventions: Drug: JNJ-0440; Drug: Placebo
- JNJ-0440 (High Dose) or Placebo (Experimental): Participants will receive single oral dose (high) of JNJ-0440 or matching placebo under fed conditions.
  Interventions: Drug: JNJ-0440; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-0440 — JNJ-0440 tablets will be administered orally.
Drug: Placebo — Matching placebo tablets will be administered orally.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of JNJ-64530440 (JNJ-0440) in healthy Japanese adult male participants after single oral dose administration with ascending dose design.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kg]/height^2 [m]^2) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 50 kilogram (kg), at time of screening
* Healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening and at admission to the study site. If the results of the biochemistry panel including liver enzymes, other specific tests, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if these are grade 1 abnormal values and the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Blood pressure (after the participants has been supine for 5 minutes) between 90 and 140 millimeter of Mercury (mm Hg) systolic, inclusive, and no higher than 90 mm Hg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 90 days after receiving the study drug

Exclusion Criteria:

* Any history of confirmed clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Clinically significant abnormal physical examination, vital signs, or 12 lead ECG at screening or at admission to the study site as deemed appropriate by the investigator
* History of confirmed clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs
* Known allergy to heparin or history of heparin induced thrombocytopenia
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as hallucinogens, barbiturates, opiates, opioids, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening or at admission to the study site

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 37 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical agent under study.
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  Cmax is defined as the maximum observed plasma analyte concentration.
Actual Sampling Time to Reach the Maximum Observed Plasma Analyte Concentration (Tmax) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  Tmax is defined as actual sampling time to reach maximum observed plasma analyte concentration.
Area Under the Plasma Concentration-time Curve from Time Zero to 24 Hours Postdose (AUC [0- 24h]) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  AUC(0-24h) is area under the plasma concentration-time curve from time zero to 24 hours, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-time Curve from Time Zero to Last Quantifiable Concentration Time (AUC [0- Last]) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  AUC(0-Last) is area under the plasma concentration-time curve from time zero to time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-time Curve from Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); where C(last) is the last observed measurable (non-below quantification limit) concentration.
Apparent Terminal Elimination Rate Constant (Lambda[z]) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent Terminal Elimination Half-Life (t1/2) of JNJ-0440 | Up to follow-up visit (approximately up to Day 9)
  The t1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic analyte concentration time curve, and is calculated as 0.693/lambda(z).
Apparent Volume of Distribution (Vdz/F) | Up to follow-up visit (approximately up to Day 9)
  The Vdz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution based on the terminal phase after extravascular administration, uncorrected for absolute bioavailability and calculated as dose/(lambda (z)*AUC[0-infinity]).
Apparent Total Clearance (CL/F) | Up to follow-up visit (approximately up to Day 9)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent total clearance of drug after extravascular administration, uncorrected for absolute bioavailability, calculated as dose/AUC(0-infinity).
Amount of JNJ-0440 Excreted in Urine within the Time Interval x to y (Ae[x-y]) | Up to 72 hours postdose
  Ae(x-y) is the amount of JNJ-0440 excreted into urine for the collection interval from x to y hours, where x and y are the start and end times of the interval, respectively, calculated by multiplying the urinary volume with the urinary concentration for that interval.
Cumulative Urinary Recovery (Ae[0-x]) | Up to 72 hours postdose
  Ae(0-x) is the sum of Ae values for all collection intervals up to 72 hours postdose.
Total Cumulative Urinary Recovery (Ae[total]) | Up to 72 hours postdose
  Ae(total) is the sum of Ae values for all collection intervals.
Percentage of JNJ-0440 Excreted in Urine (Ae%dose[0-x]) | Up to 72 hours postdose
  The Ae%dose(0-x) is the percentage of cumulative JNJ-0440 dose recovered into the urine for all collection intervals up to x hours postdose, calculated as (Ae/dose[0-x])∗100.
Percentage of JNJ-0440 Excreted in Urine (Ae%dose[total]) | Up to 72 hours postdose
  Ae%dose(total) is the percentage of total JNJ-0440 dose recovered into the urine for all collection intervals, calculated as (Ae/dose[total])∗100.
Renal Clearance (CLr) of JNJ-0440 | Up to 72 hours postdose
  The CLr is the renal clearance of the drug, calculated as Ae(total)/AUC(0-infinity).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Sumida Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency